CLINICAL TRIAL: NCT00003612
Title: Randomized Phase II Trial of Paclitaxel, Carboplatin and rhuMAb Her-2 (Herceptin) as First-Line Chemotherapy in Patients With Metastatic Breast Cancer Who Overexpress Her-2
Brief Title: Combination Chemotherapy and Trastuzumab in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-983252; CDR0000066689 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Schedule A: paclitaxel + carboplatin + trastuzumab (Experimental): Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes and then trastuzumab (Herceptin) IV over 90 minutes on day 1 of week 1. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients then receive trastuzumab IV over 30 minutes every 3 weeks until disease progression.
  Patients are followed every 3 months for 2 years and then every 6 months thereafter.
  Interventions: Biological: trastuzumab; Drug: carboplatin; Drug: paclitaxel
- Schedule B: paclitaxel + carboplatin + trastuzumab (Experimental): Patients receive paclitaxel IV over 1 hour followed by carboplatin IV over 15 minutes on day 1 of weeks 1-3 and trastuzumab IV over 90 minutes immediately after carboplatin on day 1. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive trastuzumab IV over 30 minutes every 3 weeks until disease progression.
  Patients are followed every 3 months for 2 years and then every 6 months thereafter.
  Interventions: Biological: trastuzumab; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Biological: trastuzumab
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of combining paclitaxel, carboplatin, and trastuzumab in treating women who have metastatic breast cancer that overexpresses HER2.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate associated with two different treatment schedules of paclitaxel, carboplatin, and trastuzumab (Herceptin) in women with overexpressed HER-2 growth factor receptor and metastatic breast cancer. (Schedule A closed to accrual effective 05/16/2003).
* Compare the time to progression and median survival in patients treated with these schedules.
* Compare the toxicity of these treatment schedules in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior adjuvant therapy (none vs less than 6 months vs at least 6 months), estrogen receptor (ER) status and progesterone receptor (PR) status at initial diagnosis (ER positive/PR positive or unknown vs ER positive/PR negative vs ER positive or unknown/PR negative), menopausal status (pre vs post), and performance status (0 or 1 vs 2). Patients are assigned to 1 of 2 treatment schedules.

* Schedule A: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes and then trastuzumab (Herceptin) IV over 90 minutes on day 1 of week 1. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients then receive trastuzumab IV over 30 minutes every 3 weeks until disease progression. (Schedule A closed to accrual effective 05/16/2003).
* Schedule B: Patients receive paclitaxel IV over 1 hour followed by carboplatin IV over 15 minutes on day 1 of weeks 1-3 and trastuzumab IV over 90 minutes immediately after carboplatin on day 1. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive trastuzumab IV over 30 minutes every 3 weeks until disease progression.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 36-92 patients (18-46 per treatment schedule) will be accrued for this study within 7-18.5 months. (Schedule A closed to accrual effective 05/16/2003).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the breast
* Strong overexpression of HER-2 by immunohistochemistry (3+)

  * 0-2+ tumors allowed if demonstrate amplification by FISH
* Bidimensionally measurable disease
* Brain metastasis must not represent sole site of disease
* No untreated brain metastasis receiving radiotherapy
* Previously treated brain metastases in continued response to radiotherapy and/or surgery for at least 2 months allowed
* Hormone receptor status:

  * Positive or negative

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No myocardial infarction within the past 6 months
* No congestive heart failure or unstable angina
* No clinically significant pericardial effusion or arrhythmia

Other:

* No other invasive malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No active uncontrolled infection
* No prior allergic reaction to Cremophor EL, anesthetics, or muscle relaxants
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent filgrastim (G-CSF)

Chemotherapy:

* Prior adjuvant chemotherapy allowed
* Prior taxane therapy allowed
* No prior cisplatin or carboplatin
* No prior chemotherapy for metastatic disease

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to more than 25% of marrow
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior surgery and recovered

Other:

* At least 7 days since prior parenteral antibiotics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 1999-04 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years

SECONDARY OUTCOMES:
time to progression | Up to 5 years
median survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic
Locations (25):
- United States (24):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Perez EA, Suman VJ, Rowland KM, Ingle JN, Salim M, Loprinzi CL, Flynn PJ, Mailliard JA, Kardinal CG, Krook JE, Thrower AR, Visscher DW, Jenkins RB. Two concurrent phase II trials of paclitaxel/carboplatin/trastuzumab (weekly or every-3-week schedule) as first-line therapy in women with HER2-overexpressing metastatic breast cancer: NCCTG study 983252. Clin Breast Cancer. 2005 Dec;6(5):425-32. doi: 10.3816/CBC.2005.n.047. PMID 16381626
- [Result] Perez EA, Rowland KM, Suman VJ, et al.: N98-32-52: efficacy and tolerability of two schedules of paclitaxel, carboplatin and trastuzumab in women with HER2 positive metastatic breast cancer: a North Central Cancer Treatment Group randomized phase II trial. [Abstract] Breast Cancer Res Treat 82 (Suppl 1): A-216, S47, 2003.
- [Result] Rowland KM, Suman VJ, Ingle JN, et al.: NCCTG 98-32-52: randomized phase II trial of weekly versus every 3-week administration of paclitaxel, carboplatin and trastuzumab in women with HER2 positive metastatic breast cancer (MBC). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-31, 2003.
- [Derived] Chumsri S, Sperinde J, Liu H, Gligorov J, Spano JP, Antoine M, Moreno Aspitia A, Tan W, Winslow J, Petropoulos CJ, Chenna A, Bates M, Weidler JM, Huang W, Dueck A, Perez EA. High p95HER2/HER2 Ratio Associated With Poor Outcome in Trastuzumab-Treated HER2-Positive Metastatic Breast Cancer NCCTG N0337 and NCCTG 98-32-52 (Alliance). Clin Cancer Res. 2018 Jul 1;24(13):3053-3058. doi: 10.1158/1078-0432.CCR-17-1864. Epub 2018 Mar 12. PMID 29530935